CLINICAL TRIAL: NCT06498375
Title: Fluid Status and Body Composition Analysis in Patients After Cardiac Surgery Assessed by Bioelectrical Impedance Method and Its Impact on Postoperative Morbidity and Mortality
Brief Title: Fluid Status and Body Composition Analysis by Bioelectrical Impedance in Patients After Cardiac Surgery (FLUBIACS)
Acronym: FLUBIACS
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Laura Kekec, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: TP 20230216
Record Dates: First submitted 2024-06-26; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Cardiopulmonary Disease; Fluid Overload
MeSH Terms: conditions — Pulmonary Heart Disease; Edema | interventions — Electric Impedance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On-pump cardiac surgery: Patients undergoing cardiac surgery with cardiopulmonary bypass
  Interventions: Diagnostic Test: Bioelectrical impedance
- Off-pump cardiac surgery: Patients undergoing cardiac surgery without cardiopulmonary bypass
  Interventions: Diagnostic Test: Bioelectrical impedance

INTERVENTIONS:
Diagnostic Test: Bioelectrical impedance — Fluid distribution measured by bioelectrical impedance Bodystat Multiscan 5000 Bodystat Ltd, Isle of Man, British Isles

SUMMARY:
Evaluation of fluid status in cardiac surgery patients using bioelectrical impedance and its impact on postoperative morbidity and mortality

DETAILED DESCRIPTION:
Hydration and fluid balance dynamics after cardiac surgery is complex and requires comprehensive knowledge of bluid balance dynamics. Surgical trauma, anaesthesia and use of cardiopulmonary bypass significantly influence postoperative fluid status. Deviations from normal values on the other hand can be related to increase in morbidity and mortality.

The purpose of this prospective observational clinical study is to assess fluid status using bioelectric impedance in patients undergoing cardiac surgery and to evaluate its impact on postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion criteria

1. Elective cardiovascular surgery (on-pump or off-pump)
2. Age ≥ 18 years
3. ASA 3 or 4
4. Provided verbal and written informed consent

Exclusion criteria

1. Refusal to participate in the research
2. < 18 years
3. Renal failure requiring replacement treatment with hemodialysis
4. Amputation of a limb
5. Pregnancy
6. Emergency Procedures
7. Reoperation
8. Pacemaker/implantable cardioverter-defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (18 years or over) undergoing elective cardovascular surgery (on-pump or off-pump)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Phase angle (in degrees)
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Impedance ratio
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Total body water (TBW), extracellular water (ECW), intracellular water (ICW) (in litres)
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Oedema index (ECW/TBW ratio)
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Body cell mass (in kilograms)
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Skeletal muscle mass (in kilograms)
Fluid distribution during the early postoperative period (≤ 5 days) | Perioperative period (preoperatively, on the first, third, and fifth postoperative day)
  Bioelectrical impedance vector analysis

SECONDARY OUTCOMES:
Impact of fluid distribution/fluid overload on duration of postoperative mechanical ventilation | Duration of stay in ICU (estimated to up to 5 days)
Impact of fluid distribution/fluid overload on postoperative complications (myocardial infarction, cardiogenic shock, vasoplegia, atrial fibrillation, heart failure, bleeding, infections, delirium) | Up to 1 year after the operation
Impact of fluid distribution/fluid overload on length of stay in the intensive care unit | Duration of stay in ICU (estimated to up to 5 days)
Impact of fluid distribution/fluid overload on length of hospitalisation | Duration of hospital stay (up to 1 month)
Impact of fluid distribution/fluid overload on 30-day postoperative mortality | On day 30
Impact of fluid distribution/fluid overload on 1-year postoperative mortality | At 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Taleska Štupica, MD, PhD, DESA, EDIC, Study Chair — Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre Ljubljana; Laura Kekec, MD, Principal Investigator — Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre Ljubljana; Matej Jenko, MD, Study Director — Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre Ljubljana; Maja Šoštarič, MD, PhD, Study Director — Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre Ljubljana
Locations (1):
- Department of Anaesthesiology and Surgical Intensive Care, University Medical Centre Ljubljana, Ljubljana, Slovenia